CLINICAL TRIAL: NCT03495557
Title: Evaluation of Port Site Hernia Prevalence After Prophylactic Mesh Placement Following Laparoscopic Cholecystectomy: Randomized Clinical Trial
Brief Title: Prevalence of Port Site Hernia After Mesh Placement in Laparoscopic Cholecystectomy.
Acronym: PSHERNIA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital de Mataró (Other)
Responsible Party: Principal Investigator, Ana Ciscar, MD, Hospital de Mataró
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PORT SITE HERNIA
Record Dates: First submitted 2018-03-23; First posted 2018-04-12 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Incisional Hernia
Keywords: Hernia; Cholecystectomy; Mesh fixation
MeSH Terms: conditions — Incisional Hernia; Hernia

STUDY DESIGN:
Intervention Model Description: Control will have simple closure while experimental group will have simple closure+mesh
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Sham Comparator): Simple closure
  Interventions: Procedure: Control
- Experimental (Experimental): Simple closure + mesh
  Interventions: Device: Experimental

INTERVENTIONS:
Procedure: Control — Fascial closure with simple polydioxanone suture 2/0 stitches
  Arms: Control
Device: Experimental — Onlay polypropylene mesh placement (MN mesh)
  Arms: Experimental

SUMMARY:
A prophylactic mesh fixation after fascial closure in umbilical trocar after cholecystectomy may prevent the trocar site hernia incidence. Especially in patients who present certain risk factors.

DETAILED DESCRIPTION:
Randomized controlled trial. Patients with more than two incisional hernia risk factors (age ≥70, BMI ≥30, diabetes mellitus, fascial enlargement) who undergo elective/emergent cholecystectomy. Control arm: fascial closure with simple PDS 2/0 Stitches. Study arm: fascial closure with simple PDS 2/0 stitches and onlay polypropylene mesh placement. Main outcome umbilical trocar site hernia incidence during a 3 years follow up. Clinical and radiological assessment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Laparoscopic cholecystectomy
* Emergent/elective
* ≥2 risk factors: diabetes mellitus, age ≥70 years, BMI ≥30, fascial enlargement

Exclusion Criteria:

* Conversion to laparotomy
* Emergent re intervention
* Immunosuppression
* Umbilical hernia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Umbilical trocar site hernia incidence | 3 years
  Umbilical trocar site hernia incidence after 6 months and 1 year (clinical assessment) and after 3 years (radiological confirmation)

SECONDARY OUTCOMES:
Seroma incidence | 6 months
  A mass or tumefaction caused by the localized accumulation of serum within the tissue (clinical assessment)
Hematoma incidence | 6 months
  A localized collection of extravasated blood clotted under the tissue (clinical assessment)
Wound infection incidence | 6 months
  Combination of redness, swelling, warm and/or fluid drainage in the wound assessed clinically
Pain presence | 6 months, 1 and 3 years
  Pain presence related to the umbilical wound scored from 0 (no pain) to 10 (severe pain)
Hospital discharge | 48 hours
  When patients leave the hospital after the intervention, measured by hours
Operative time | 2 hours
  Intervention duration, measured by minutes
Return to regular activity | 6 months
  When patient return to job or regular activities after surgery, measured by days
Patient satisfaction | 3 years
  How satisfied/unsatisfied is the patient with the whole process measured by a survey form which classify it in a range from 0 (very unsatisfied) to 5 (very satisfied)
Surgeon satisfaction | 3 years
  How satisfied/unsatisfied is the surgeon with the whole process measured by a survey form which classify it in a range from 0 (very unsatisfied) to 5 (very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Ciscar, MD, Principal Investigator — Hospital de Mataró
Locations (1):
- Hospital de Mataró, Mataró, Barcelona, Spain

REFERENCES:
- [Derived] Ciscar A, Sanchez-Saez E, Vila Tura M, Ruiz de Leon P, Gomez Pallares M, Troyano Escribano D, Abadal Prades M, Mans Muntwyler E, Pereira JA, Badia JM. Assessment of the effectiveness of a polypropylene onlay mesh in the prevention of laparoscopic trocar-site incisional hernia in high-risk patients. A randomized clinical trial. Hernia. 2024 Dec;28(6):2187-2194. doi: 10.1007/s10029-024-03124-7. Epub 2024 Aug 29. PMID 39207550